CLINICAL TRIAL: NCT01095991
Title: A Randomised, Open, Phase I Study in Patients With Type 2 Diabetes Mellitus Treated With Metformin to Evaluate the Effect of AZD1656 on the Pharmacokinetics of Sitagliptin and Vice Versa
Brief Title: Investigate the Effect of AZD1656 on the Pharmacokinetics of Sitagliptin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00032
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, Sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD1656, day 1-5, AZD1656 + Sitagliptin day 6-10, Sitagliptin day 11-15.
  Interventions: Drug: AZD1656; Drug: Sitagliptin
- 2 (Experimental): Sitagliptin day 1-5, AZD1656 + Sitagliptin day 6-10, AZD1656 day 11-15.
  Interventions: Drug: AZD1656; Drug: Sitagliptin

INTERVENTIONS:
Drug: AZD1656 — Oral tablet bd,
Drug: Sitagliptin — Oral tablet od
  Other Names: Januvia

SUMMARY:
The purpose of this study is to evaluate the effects of AZD1656 on Sitagliptin pharmacokinetics and vice versa in patients with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed type 2 diabetes mellitus for at least 2 months and treated with metformin.
* Body mass index between ≥19 and ≤42 kg/m2.

Exclusion Criteria:

* Intake of another investigational drug within the last 30 days prior to enrolment.
* Clinically significant illness or clinically relevant trauma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of AZD1656 on the steady-state PK of sitagliptin and vice versa by assessment of AUC0-24 and Cmax | Serial PK sampling will be done on Days 5, 10 and 15

SECONDARY OUTCOMES:
To evaluate the effect of AZD1656 on the steady-state PK of sitagliptin and vice versa by assessment of tmax, t1/2 and CL/F | Serial PK sampling will be done on Days 5, 10 and 15
To evaluate the PK of the AZD1656 and its metabolite when AZD1656 is administered with and without sitagliptin by assessment of AUC0-24, Cmax, tmax and t1/2 | Serial PK sampling will be done on Days 5, 10 and 15
To evaluate the safety of AZD1656 with and without sitagliptin by assessment of adverse events (AEs), physical examination, electrocardiogram (ECG), pulse, blood pressure (BP), weight and FPG. | Paper ECG (days 1,2,3,6,7,8,11,16), BP/pulse preentry, every residential day. Weight, physical examination preentry and follow-up. FPG on preentry, day 1,6 and 11.

CONTACTS AND LOCATIONS:
Overall Officials: Stanko Skrtic, Study Director — AstraZeneca Molndal Sweden; Christoph Kapitza, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH; Mirjana Kujacic, Study Director — AstraZeneca Molndal Sweden
Locations (1):
- Research Site, Neuss, Germany